CLINICAL TRIAL: NCT04858256
Title: Phase 2, Open Label, Multicenter Study of Pacritinib in Relapsed/Refractory T-cell Lymphoproliferative Neoplasms
Brief Title: Pacritinib in Relapsed/Refractory T-cell Lymphoproliferative Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Hoosier Cancer Research Network (Other); CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2020.064; R01CA265929 (NIH); HUM00184365 (Other: University of Michigan); HCRN LYM21-544 (Other: Hoosier Cancer Research Network)
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: T-Cell Neoplasm; Lymphoproliferative Disorders
Keywords: pacritinib
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Intervention Model Description: Each of the four disease-based cohorts will be run in parallel, independently, and under an identical two-stage design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: PTCL, NOS (Experimental): Patients will receive single agent pacritinib.
  Interventions: Drug: Pacritinib
- Cohort 2: AITL/TFH PTCL (Experimental): Patients will receive single agent pacritinib.
  Interventions: Drug: Pacritinib
- Cohort 3: CTCL (MF/SS) (Experimental): Patients will receive single agent pacritinib.
  Interventions: Drug: Pacritinib
- Cohort 4: Less common PTCL subtypes (Experimental): Patients will receive single agent pacritinib.
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Pacritinib will be dosed at 200mg twice daily.

SUMMARY:
The main purpose of this study is to determine the effectiveness of the study drug pacritinib in people with relapsed or refractory lymphoproliferative disorders.

DETAILED DESCRIPTION:
Patients will receive single-agent treatment with pacritinib 200mg orally twice daily until any condition for treatment discontinuation has been met. Patients will be enrolled into one of four cohorts: Peripheral T-Cell Lymphoma, not otherwise specified (PTCL, NOS) (cohort 1); angioimmunoblastic T-cell lymphoma/follicular helper T-cell (AITL/TFH) PTCL (cohort 2); Cutaneous T-Cell Lymphoma (CTCL) - mycosis fungoides (MF) and Sezary syndrome (SS) (cohort 3); and other eligible, less common PTCL subtypes (cohort 4).

14NOV2025- Updates were made to the inclusion and exclusion criteria to align with the pacritinib IB v19 and the funders guidance.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately. Subject must have the ability to understand and the willingness to sign a written informed consent.
2. ECOG performance status ≤ 2
3. A histologically confirmed diagnosis, per the WHO 2016 classification, of any PTCL or CTCL subtype listed in the protocol.
4. Relapsed or refractory disease. Refractory disease is defined as progression during treatment or recurrent/progressive disease within 6 months of completing a treatment regimen that achieved either stable disease or a PR/CR. Relapsed disease is defined as progression or recurrence at least 6 months after a prior documented response (PR or CR).
5. Adequate organ and hematopoietic function as defined in the protocol.
6. Sufficient archival tissue (15 unstained slides obtained within 90 days prior to registration) is required. If available, this tissue should be identified at screening and shipped prior to C2D1.If not available, a lymph node or tissue biopsy (core-needle or excisional) or skin biopsy (for CTCL) is required. The type of tissue obtained is at the discretion of the investigator based on disease. NOTE: If archival tissue is not available and a fresh biopsy is inaccessible or technically challenging (per site investigator discretion) at the site, the subject may be eligible for the study.
7. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Testing is based on known history and local policies.
8. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. Testing is based on known history and local policies.
9. Ability to take oral medication without crushing, dissolving or chewing tablets.
10. In the investigator's opinion, the patient requires treatment, has an anticipated life expectancy of at least 3 months, and the patient has the ability to communicate satisfactorily with the investigator and the study team, to participate fully in the study, and comply with all requirements.

Selected Exclusion Criteria:

1. History of, or a concurrent, clinically significant illness, medical condition or laboratory abnormality that, in the investigator's opinion, could affect the conduct of the study
2. Pregnant or breast feeding women. NOTE: women may not breast feed or store breast milk during treatment and for 3 months after pacritinib discontinuation.
3. Unwilling or unable to use a medically acceptable form of contraception during the time of participation in the trial (sexual abstinence is permissible) unless documented successful vasectomy, hysterectomy, bilateral oophorectomy or post-menopausal for at least 2 years. Women of childbearing potential must use highly effective methods of birth control from the time of informed consent, for the duration of pacritinib treatment and for 30 days after discontinuation of pacritinib. This timeframe also applies to breast-feeding and egg donation. Fertile males must use contraception from the time of study treatment initiation, for the duration of pacritinib treatment and for 30 days after discontinuation of pacritinib. This timeframe is also applicable to sperm donation. Participants should be informed of the risk of unintended pregnancy due to potential reduced effectiveness of hormonal contraceptives sensitive to CYP3A4 metabolism (i.e. progestin) during treatment with pacritinib.
4. Uncontrolled current illness, including, but not limited to the following:

   1. Ongoing or active infections requiring intravenous antimicrobials
   2. Symptomatic congestive heart failure (CHF) defined as NYHA class II, III or IV (Appendix II), or ejection fraction <45% in any patient.
   3. Unstable angina pectoris within 6 months of study enrollment
   4. Unstable cardiac arrhythmia
   5. History of myocardial infarction, stroke or intracranial hemorrhage within 6 months prior to enrollment
   6. Moderate to severe hepatic impairment (Child-Pugh class B or C).
   7. Psychiatric illness or social situations that would limit compliance with study requirements.
5. Recent (within 21 days of initiation of therapy, day 1) major surgery
6. Less than 14 days have elapsed since last radiation therapy or chemotherapy treatment or patient has not recovered from all clinically significant treatment related toxicity; less than 90 days have passed since date of autologous stem cell transplant and patient has not recovered to ≤grade 1 toxicity related to this procedure.
7. Use of systemic steroids at a dose equivalent to >10 mg/day of prednisone
8. Prior treatment with pacritinib
9. Requires use of a medication that increases the risk of bleeding, including anticoagulation or antiplatelet therapy with the exception of aspirin at doses of ≤ 100mg daily.
10. History of significant bleeding (≥ Grade 2 by CTCAE), bleeding diatheses, or bleeding complications within the past 3 months.
11. Hypersensitivity or allergic reaction to compounds related to pacritinib.
12. Treatment with strong CYP3A4 inducers or strong CYP3A4 inhibitors (See Appendix III), for which no alternative is available. Treatment with strong CYP3A4 inducers or strong CYP3A4 inhibitors requires a washout period of 2 weeks prior to initiation of therapy, Cycle 1 Day 1.
13. Uncontrolled diarrhea. NOTE: patients with chronic diarrhea that is well controlled with supportive care measure (e.g. anti-motility agents) are eligible
14. Any gastrointestinal or metabolic condition that in the opinion of the investigator could interfere with the absorption of an oral medication.
15. Prior allogeneic stem-cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  ORR will be estimated for each disease-specific cohort of patients. Overall response is defined as best disease response recorded from first day of treatment until disease progression or treatment discontinuation. Response in PTCL patients is assessed by PET/CT scan using the Response Evaluation Criteria in Lymphoma (RECIL) criteria. Response in CTCL patients is assessed using the modified Severity Weighted Assessment Tool (mSWAT). Results will be stratified by type: complete response [CR], partial response [PR], minor response [MR; a provisional category in RECIL only], stable disease [SD], progressive disease [PD]; and by cohort.

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to approximately 5 years
  CRR is defined as the percentage of PTCL patients who have a best response of CR per the RECIL criteria and percentage of CTCL who a have a best response of CR per the modified Severity Weighted Assessment Tool (mSWAT). CR rate will be analyzed by cohort and summarized with "time-to-event" analysis.
Duration of response (DOR) | Up to approximately 5 years
  DOR is defined as time from first observed response (CR or PR) to date of progression (PD) or death, whichever occurs first. DOR will be analyzed by cohort with "time-to-event" analysis.
Time to next treatment (TTNT) | Up to approximately 5 years
  TTNT is defined as time from first dose of pacritinib to initiation of alternative systemic, antineoplastic therapy. TTNT will be analyzed by cohort using a "time-to-event" analysis.
Progression- free survival (PFS). | Up to approximately 5 years
  PFS is defined as the time from first day of treatment to date of disease progression (PD) or death, whichever occurs first. Patients who survive without progression will be censored on the date of last evaluable tumor assessment. PFS will be analyzed by cohort and summarized with "time-to-event analysis.
Treatment related toxicities >=grade 3 | 30 days post end of treatment (+4 days)
  The analyses of safety endpoint will be conducted using tabulations of adverse events, assessed per NCI CTCAE v5.0, stratified by grade (severity) and attribution for each cohort. Grade 3 or higher treatment related toxicities will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Wilcox, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Duke Cancer Institute, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No